CLINICAL TRIAL: NCT06903377
Title: A Multicenter, Open-label, Dose-Escalation and Dose-Expansion Phase I/II Study of ZG005 Combined With Gecacitinib in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Study of ZG005 Combined With Gecacitinib in Patients With Advanced Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZG005-JAK-001
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part1-Group A (Experimental): ZG005 20mg/kg IV Q3W+Gecacitinib 50mg po Bid
  Interventions: Biological: ZG005 for Injection; Drug: Gecacitinib Hydrochloride Tablets
- Part1-Group B (Experimental): ZG005 20mg/kg Q3W+Gecacitinib 100mg po Bid
  Interventions: Biological: ZG005 for Injection; Drug: Gecacitinib Hydrochloride Tablets

INTERVENTIONS:
Biological: ZG005 for Injection — intravenous infusion
  Other Names: ZG005
Drug: Gecacitinib Hydrochloride Tablets — Oral
  Other Names: Gecacitinib

SUMMARY:
This is a multicenter Phase I/II study for patients with advanced non-small cell lung cancer who have failed PD-1/L1 therapy, aiming to evaluate the safety of ZG005 in combination with Gecacitinib in this population, as well as the preliminary efficacy of this combination regimen.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand this study and voluntarily sign the ICF.
* Age 18-75 years, no gender restriction.
* Patients with locally advanced or recurrent/metastatic squamous and/or non-squamous non-small cell lung cancer confirmed by histology/cytology, unsuitable for radical therapy.

Exclusion Criteria:

* Medical history, CT scan, or MRI indicates the presence of CNS metastases.
* Other malignancies within 5 years.
* Any other reason deeming the participant unsuitable for the study, as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Adverse Event (AE) | Up to 2 years

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China